CLINICAL TRIAL: NCT00644072
Title: Phase I Study of SNX-5422 Mesylate in Adults With Refractory Solid Tumor Malignancies and Lymphomas
Brief Title: SNX-5422 to Treat Solid Tumor Cancers and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080091; 08-C-0091
Record Dates: First submitted 2008-03-25; First posted 2008-03-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-06-16

CONDITIONS: Lymphoma; Neoplasms
Keywords: Hsp90 Inhibitor; Her2; Neoplasms; Advanced Cancer; Cancer; Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma; Neoplasms | interventions — SNX-5422

INTERVENTIONS:
Drug: SNX-5422

SUMMARY:
Background:

SNX-5422 is an experimental drug that inhibits a protein called Hsp90, which is important for the growth of tumor cells.

SNX-5422 has shown some activity against tumors in the laboratory and animal studies.

Objectives:

To determine the highest safe dose, or maximum tolerated dose (MTD), of SNX-5422 that can safely be given to patients with solid tumor cancers and lymphomas when taken twice a week.

To learn how the body's blood and tissue cells react to SNX-5422.

To examine the effects of SNX-5422 on tumors and lymphomas.

Eligibility:

Patients 18 years of age or older who have solid tumor cancers or lymphomas that do not respond to standard therapy or for whom no acceptable standard treatment is available.

Design:

SNX-5422 is taken by mouth twice a week in 28-day cycles. Treatment may continue as long as the cancer does not worsen and side effects are acceptable. Three to six patients are enrolled in the study at a time. Each group is given a higher dose of SNX-5422 than the previous, as long as the preceding dose was tolerated and until the MTD is determined. When the MTD is found, six more patients are enrolled at that dose level.

During the treatment period, patients undergo the following tests and procedures:

* Clinic visits for a physical examination each treatment cycle to check on health status.
* Blood tests for routine laboratory values, to determine how the body handles SNX-5422, and to examine the effects of SNX-5422 on blood cells and other targets.
* Urine tests as needed, depending on the results of blood tests.
* CT scans, or other imaging tests every 8 weeks to evaluate the tumor response to treatment.
* Tumor biopsy (surgical removal of a tissue sample for examination under a microscope) before the first dose of SNX-5422 and again 24 hours after the first dose to see how the drug affects the tumor. This test is optional.

DETAILED DESCRIPTION:
Background:

* Inhibitors of the chaperone protein Hsp90 are of current interest because of the central role that Hsp90 plays in the maturation and maintenance of numerous proteins, such as Her2, critical for tumor cell viability and growth.
* Disruption of Hsp90 function has been shown to cause degradation of multiple Hsp90 client proteins, leading to inhibition of several key signaling pathways. This in turn results in inhibition of cellular proliferation.

Objectives:

* Determine the maximum tolerated dose (MTD) of SNX-5422 when administered twice a week for 28 days.
* Characterize the safety profile of SNX-5422 when administered twice a week for 28 days.
* Investigate the effects of SNX-5422 on Hsp90 client proteins using pharmacodynamic (PD) assays.
* Investigate the effects of SNX-5422 on tumor and lymphoma response using the National Cancer Institute (NCI) Response Evaluation Criteria in Solid Tumors (RECIST) criteria) and standardized lymphoma criteria, respectively.
* Determine the pharmacokinetic (PK) profile of SNX-2112 and its prodrug SNX-5422 in humans.

Eligibility:

* Patients with histologically documented solid tumors and lymphoid malignancies (lymphoma and CLL) whose disease has progressed following standard therapy, or who have no acceptable standard treatment options.
* Patients with no major surgery, radiation, or chemotherapy within 4 weeks prior to study enrollment, and who have recovered from toxicities from prior therapies to at least eligibility levels.

Design:

This will be a Phase I dose escalation study to determine the MTD and recommended Phase II dose of SNX-5422. SNX-5422 will be administered orally twice a week for 28 days in continuous cycles until disease progression occurs or the patient meets off-study criteria. Three to six patients will be enrolled at each dose level, and up to 6 additional patients at the MTD, for a minimum of up to 36 patients and a maximum of 60 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with histologically documented (by the NIH pathology department) solid tumors and lymphoid malignancies (lymphoma and CLL) who are refractory to standard therapy or who have no acceptable standard treatment options. Patients with lymphoid malignancies will be eligible if their disease has progressed following 2 standard therapies (aggressive NHL), and if their disease is considered refractory (for indolent NHL).

Patients must have measurable or evaluable disease.

Patients must have recovered to at least Grade less than or equal to1 toxicity levels due to adverse events and/or toxicity of prior chemotherapy or biologic therapy. They must not have had chemotherapy or biologic therapy within 4 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin C, or UCN-01). Patients must be greater than or equal to 2 weeks since any prior administration of study drug in an exploratory IND/Phase Zero study. Patients must be greater than or equal to 1 month since any prior radiation or major surgery. However, patients receiving bisphosphonates for any cancer or undergoing androgen deprivation therapy for prostate cancer are eligible for this therapy.

Age greater than or equal to 18 years

The Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).

Life expectancy greater than 3 months

Patients must have normal or adequate organ and marrow function as defined below:

* Absolute neutrophil count greater than or equal to 1,500/milliliter
* Platelets greater than or equal to 100,000/milliliter
* Total bilirubin* within less than or equal to 1.5 times upper limit of normal
* AST (SGOT)/ALT (SGPT) less than or equal to 2.5 times institutional upper limit of normal
* creatinine less than 1.5 times upper limit of normal

OR

- creatinine clearance greater than or equal to 60 mL/min (measured) for patients with creatinine levels greater than or equal to 1.5 times upper limit of normal.

*we will allow patients with Gilbert's syndrome with total bilirubin up to 2.5 mg/dL

The effects of SNX-5422 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry, for the duration of study participation, and for 2 months after discontinuation from the study. Women of childbearing potential must have a negative pregnancy test in order to be eligible. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SNX-5422, breastfeeding should be discontinued if the mother is treated with SNX-5422.

Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Patients receiving any other investigational agents. Patients with symptomatic brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, patients who have had treatment for their brain metastases and whose brain metastatic disease status has remained stable for at least 3 months without steroids may be enrolled at the discretion of the principal investigator.

Uncontrolled medical illness including, but not limited to, ongoing or uncontrolled, symptomatic congestive heart failure (AHA Class II or worse), uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

HIV-positive patients receiving combination antiretroviral therapy are excluded from the study because of possible PK interactions with SNX-5422. HIV positive patients not receiving antiretroviral therapy are excluded due to the possibility that SNX-5422 may worsen their condition and the likelihood that the underlying condition may obscure the attribution of adverse events with respect to SNX-5422.

Chronic diarrhea.

Gastrointestinal diseases that could affect drug absorption, including postsurgical states such as gastric bypass.

Gastrointestinal diseases that could alter the assessment of safety, including irritable bowel syndrome, ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-03-07; Primary Completion 2009-06-30 (Actual); Study Completion 2011-06-16 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of SNX-5422 when administered twice a week for 28 days.

SECONDARY OUTCOMES:
Investigate the effects of SNX-5422 on Hsp90 client proteins using pharmacodynamic (PD) assays.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chung EJ, Lee MJ, Lee S, Trepel JB. Assays for pharmacodynamic analysis of histone deacetylase inhibitors. Expert Opin Drug Metab Toxicol. 2006 Apr;2(2):213-30. doi: 10.1517/17425255.2.2.213. PMID 16866608
- [Background] Chung EJ, Lee S, Sausville EA, Ryan Q, Karp JE, Gojo I, Telford WG, Lee MJ, Kong HS, Trepel JB. Histone deacetylase inhibitor pharmacodynamic analysis by multiparameter flow cytometry. Ann Clin Lab Sci. 2005 Autumn;35(4):397-406. PMID 16254255
- [Background] Posadas EM, Gulley J, Arlen PM, Trout A, Parnes HL, Wright J, Lee MJ, Chung EJ, Trepel JB, Sparreboom A, Chen C, Jones E, Steinberg SM, Daniels A, Figg WD, Dahut WL. A phase II study of perifosine in androgen independent prostate cancer. Cancer Biol Ther. 2005 Oct;4(10):1133-7. doi: 10.4161/cbt.4.10.2064. Epub 2005 Oct 1. PMID 16138006